CLINICAL TRIAL: NCT04774939
Title: FinnTrunk, EVLA and Optimal Timing of Sclerotherapy
Brief Title: EVLA and Optimal Timing of Sclerotherapy
Acronym: FinnTrunk
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Central Hospital (Other); Oulu University Hospital (Other); Tampere University Hospital (Other); Päijänne Tavastia Central Hospital (Other); Satasairaala (Other); Vaasa Central Hospital, Vaasa, Finland (Other)
Responsible Party: Principal Investigator, Khalil Firoozi, MD, Turku University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 93 /1801/2020
Record Dates: First submitted 2021-02-24; First posted 2021-03-01 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Venous Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EVLA only (Active Comparator): Only main trunk/trunks with venous reflux will be treated
  Interventions: Procedure: Endovenous laser ablation
- EVLA and sclerotherapy of tributaries (Active Comparator): Main trunk/trunks with venous reflux will be treated combined with foam sclerotherapy
  Interventions: Procedure: Endovenous laser ablation

INTERVENTIONS:
Procedure: Endovenous laser ablation — The aim is to combine the significance of for sclerotherapy at the primary EVLA treatment
  Other Names: Endovenous laser ablation combined with foam sclerotherapy of varicose tributaries

SUMMARY:
The aim of the study is to investigate the optimal timing of sclerotherapy for treatment of varicose tributaries on EVLA (endogenous laser ablation) patients.

DETAILED DESCRIPTION:
The study inclusion criteria is patients with main trunk (VSM, SSV, AASV) reflux to be treated with EVLA, suffering C2-C3 varicose disease, age 18-years and no severe co-morbidities.

Patients with written consent will be randomized to two primary treatments groups; EVLA only and EVLA combined with sclerotherapy of varicose tributaries. The primary outcome is the requirement additional sclerotherapy on 3 month control visit. Other study outcomes are pain, quality of life (veins questionnaire), severity score and also recurring of varicose disease at 1, 3 and 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Varicose disease of lower extremity caused by reflux of VSM, SSV or AASV to be treated with EVLA. Age over 18 years. Clinical symptoms C2-3.

Exclusion Criteria:

* No severe comorbidities. Previous DVT.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-03-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2030-03-15 (Estimated)

PRIMARY OUTCOMES:
re-intervention | 3 months
  Requirement of re-intervention
Pain after procedure | up to 3 months after the treatment
  Post procedural pain measured with VAS scale
Quality of life before after procedure | up to 5 years
  Quality of life will be measured with Veins questionnaire
Recur | up to 5 years
  The recurring varicose veins

SECONDARY OUTCOMES:
Surgical complications | 3 months
  Infections, DVT, Pulmonary embolus will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Harri Hakovirta, Professor, Study Chair — University of Turku
Locations (1):
- Turku University Hospital, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Viljamaa J, Firoozi K, Venermo M, Pokela M, Pihlaja T, Halmesmaki K, Hakovirta H. A study protocol for comparing the treatment of varicose tributaries either concomitantly with or separately from endovenous laser ablation of the incompetent saphenous trunk (the FinnTrunk Study). A multicenter parallel-group randomized controlled study. PLoS One. 2023 May 23;18(5):e0285823. doi: 10.1371/journal.pone.0285823. eCollection 2023. PMID 37220130